CLINICAL TRIAL: NCT02629432
Title: Image-Based Structural and Functional Phenotyping of the COSYCONET Cohort Using MRI and CT (MR COPD)
Brief Title: Image-Based Structural and Functional Phenotyping of the COSYCONET Cohort Using MRI and CT
Acronym: MR-COPD
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Philipps University Marburg (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Biederer, Prof. Dr., University Hospital Heidelberg
Other Study IDs: 01GI0884
Record Dates: First submitted 2015-10-23; First posted 2015-12-14 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: MRI; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cosyconet COPD Cohort: MRI and CT of the lung will be performed in a multi-centre cohort of 625 COPD-patients from the main COSYCONET cohort.

SUMMARY:
The main objective of this trial is to prove that MRI - as the imaging modality without the use of ionizing radiation - can replace CT for structural and functional regional phenotyping of COPD. The identification of different COPD phenotypes, such as the "emphysema-type" and the "airway-type", is important because therapy and prognosis will be different. The medical problem addressed in this trial is the image-based phenotyping of COPD. The sensitivity and specificity of MRI will be compared to Lowdose-CT serving as the gold standard. MRI and CT of the lung will be performed in a multi-centre cohort of 625 COPD-patients from the main COSYCONET cohort. The reliability of the MRI results will be demonstrated. MRI phenotypes will be evaluated visually and using software with quantitative read-outs. The agreement of both will be determined. The additional information of MRI over CT will be assessed.

DETAILED DESCRIPTION:
This prospective trial aims to phenotype COPD by using Imaging methods.The identification of different COPD phenotypes, such as the "emphysema-type" and the "airway-type", is important because therapy and prognosis will be different. Imaging might play a central role in diagnosing these phenotypes. So far computed tomography (CT) is regarded as the gold standard, but it involves ionizing radiation and lacks functional information. The medical problem addressed in this trial is the image-based phenotyping of COPD. The principal research question is whether magnetic resonance imaging (MRI) can replace CT for the characterization of COPD by "structural and functional phenotyping" on a regional basis. The sensitivity and specificity of MRI will be compared to CT serving as the gold standard. To achieve this goal, MRI and CT of the lung will be performed in a multi-centre cohort of 625 COPD-patients from the main Cosyconet cohort. Also, the reliability of the MRI results will be demonstrated. MRI phenotypes will be evaluated visually and using software with quantitative read-outs. The agreement of both will be determined. The additional information of MRI over CT will be assessed. A special focus will be to implement an image-based biomarker of pulmonary functional reserve derived from the MRI measurement of pulmonary perfusion, which will be correlated with results from pulmonary functions tests (e.g. the lung transfer factor for carbon monoxide (TLCO)) the 6-minute walking test (6-MWD), and extrapulmonary disease manifestations.

ELIGIBILITY:
Inclusion Criteria:

* The population to be studied is determined by the main Cosyconet-cohort.

Key inclusion criteria:

* being included into the main cohort
* diagnosis of COPD (GOLD criteria)
* availability for repeated study visits
* male or female
* age > 40 years

Exclusion Criteria:

* Key exclusion criteria as determined by the main Cosyconet-cohort:
* having undergone lung surgery (e.g., lung volume reduction, lung transplant)
* moderate or severe exacerbation within the last 4 weeks prior to visit 1
* unable to understand the intention of the project
* lack of signed patient informed consent
* contraindications for MRI
* pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This Trial is fully embedded within the main cohort of the Cosyconet-Study: Impact of Systemic Manifestations/Comorbidities on Clinical State, Prognosis, Utilisation of Health care Ressources in Patients with COPD (COSYCONET), NCT01245933 ). Only patients included into the main study are asked to take part in this sub-trial which is not pharmaceutical and only has one arm including the expected number of patients (625) .
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of MRI for the diagnosis of emphysema-predominant vs. airway-predominant COPD phenotype based on semi-quantitative visual image evaluation with CT as standard of reference | single time point/baseline only
  diagnostic study, MRI and CT acquired on the same day

SECONDARY OUTCOMES:
number of completed examinations with diagnostic image quality to determine the achievable diagnostic quality of lung MRI in a multi-center setting | single time point/baseline only
  to assess the achievable image quality in a multicentre setting
agreement of visual and software-based phenotyping on MRI and CT (airway wall thickening, air trapping, emphysema, lung perfusion deficits) | single time point/baseline only
  to compare both modalities for the assessment of those parameters
correlation of MRI metrics with clinical tests: predictive value of perfusion MRI for pulmonary functional reserve compared to clinical tests, i.e. pulmonary function tests (TLCO) and six-minute walk test (6 MWT) | single time point/baseline only
  to assess the value of MRI-based biomarkers in comparison to clinical data
number of cases in which MRI (i.e. functional parameters) produces clinically relevant additional information to CT | single time point/baseline only
  to assess potential advantages of MR compared to CT

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Biederer, Professor, Principal Investigator — University Hospital Heidelberg; Bertram Jobst, Dr., Principal Investigator — University Hospital Heidelberg
Locations (15):
- Germany (15):
  - Universitätsklinikum, Diagnostische und Interventionelle Radiologie und Neuroradiologie, Essen
  - Universitätsklinikum Gießen und Marburg GmbH,Klinik für Diagnostische und Interventionelle Radiologie, Giessen
  - Universitätsmedizin Greifswald, Institut für Diagnostische Radiologie u. Neuroradiologie, Greifswald
  - LungenClinic Grosshansdorf, Pneumologisches Forschungsinstitut, Großhansdorf
  - Hamburger Institut für Therapieforschung (HIT) GmbH, Hamburg
  - Medizinische Hochschule Hannover, Zentrum Radiologie, Institut für Diagnostische und Interventionelle Radiologie, Hanover
  - Universitätsklinikum Heidelberg, Diagnostische und Interventionelle Radiologie, Heidelberg
  - Thoraxklinik Heidelberg, Diagnostische und Interventionelle Radiologie, Heidelberg
  - Universitätsklinikum des Saarlandes, Klinik für Diagnostische und Interventionelle Radiologie, Homburg
  - Universitätsklinikum Schleswig Holstein, Klinik für Diagnostische Radiologie, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Department für Bildgebung und Strahlenmedizin, Leipzig
  - Universitätsklinikum, Zentrum für Radiologie, Klinik für Diagnostische und Interventionelle Radiologie, Marburg
  - Institut für Klinische Radiologie, Klinikum der Universität Muenchen (KUM), Campus Innenstadt Muenchen, München
  - Klinikum der Universität Muenchen, Institut für Klinische Radiologie, München
  - Klinikum Nord-Nuernberg, Radiologie, Nuremberg

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized Data from structured image reads will be transferred to the central COSYCONET data bank in Hannover. Application form for project proposals and data retrieval can be downloaded here: http://www.asconet.net/html/cosyconet/projects?clps4835_49326291=1

REFERENCES:
- [Background] Biederer J, Mirsadraee S, Beer M, Molinari F, Hintze C, Bauman G, Both M, Van Beek EJ, Wild J, Puderbach M. MRI of the lung (3/3)-current applications and future perspectives. Insights Imaging. 2012 Aug;3(4):373-86. doi: 10.1007/s13244-011-0142-z. Epub 2012 Jan 15. PMID 22695943
- [Background] Biederer J, Beer M, Hirsch W, Wild J, Fabel M, Puderbach M, Van Beek EJ. MRI of the lung (2/3). Why ... when ... how? Insights Imaging. 2012 Aug;3(4):355-71. doi: 10.1007/s13244-011-0146-8. Epub 2012 Feb 13. PMID 22695944
- [Background] Wild JM, Marshall H, Bock M, Schad LR, Jakob PM, Puderbach M, Molinari F, Van Beek EJ, Biederer J. MRI of the lung (1/3): methods. Insights Imaging. 2012 Aug;3(4):345-53. doi: 10.1007/s13244-012-0176-x. Epub 2012 Jun 13. PMID 22695952
- [Background] Eichinger M, Optazaite DE, Kopp-Schneider A, Hintze C, Biederer J, Niemann A, Mall MA, Wielputz MO, Kauczor HU, Puderbach M. Morphologic and functional scoring of cystic fibrosis lung disease using MRI. Eur J Radiol. 2012 Jun;81(6):1321-9. doi: 10.1016/j.ejrad.2011.02.045. Epub 2011 Mar 23. PMID 21429685
- [Background] COPDGene CT Workshop Group; Barr RG, Berkowitz EA, Bigazzi F, Bode F, Bon J, Bowler RP, Chiles C, Crapo JD, Criner GJ, Curtis JL, Dass C, Dirksen A, Dransfield MT, Edula G, Erikkson L, Friedlander A, Galperin-Aizenberg M, Gefter WB, Gierada DS, Grenier PA, Goldin J, Han MK, Hanania NA, Hansel NN, Jacobson FL, Kauczor HU, Kinnula VL, Lipson DA, Lynch DA, MacNee W, Make BJ, Mamary AJ, Mann H, Marchetti N, Mascalchi M, McLennan G, Murphy JR, Naidich D, Nath H, Newell JD Jr, Pistolesi M, Regan EA, Reilly JJ, Sandhaus R, Schroeder JD, Sciurba F, Shaker S, Sharafkhaneh A, Silverman EK, Steiner RM, Strange C, Sverzellati N, Tashjian JH, van Beek EJ, Washington L, Washko GR, Westney G, Wood SA, Woodruff PG. A combined pulmonary-radiology workshop for visual evaluation of COPD: study design, chest CT findings and concordance with quantitative evaluation. COPD. 2012 Apr;9(2):151-9. doi: 10.3109/15412555.2012.654923. Epub 2012 Mar 19. PMID 22429093
- [Background] Gietema HA, Muller NL, Fauerbach PV, Sharma S, Edwards LD, Camp PG, Coxson HO; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) investigators. Quantifying the extent of emphysema: factors associated with radiologists' estimations and quantitative indices of emphysema severity using the ECLIPSE cohort. Acad Radiol. 2011 Jun;18(6):661-71. doi: 10.1016/j.acra.2011.01.011. Epub 2011 Mar 9. PMID 21393027